CLINICAL TRIAL: NCT03410901
Title: Intratumoral Injection of SD-101, an Immunostimulatory CpG, in Combination With BMS-986178 and Local Radiation in Low-Grade B-Cell Lymphomas
Brief Title: TLR9 Agonist SD-101, Anti-OX40 Antibody BMS 986178, and Radiation Therapy in Treating Patients With Low-Grade B-Cell Non-Hodgkin Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ronald Levy (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Ronald Levy, Robert K. and Helen K. Summy Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-44250; NCI-2017-02452 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LYMNHL0144 (Other: OnCore); R35CA197353 (NIH)
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: B-Cell Non-Hodgkin Lymphoma; Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3a Follicular Lymphoma; Lymphoplasmacytic Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (radiation therapy, SD-101, BMS-986178) (Experimental): Patients receive radiation therapy on days 1-2, TLR9 agonist SD-101 and anti-OX40 antibody BMS-986178 intratumorally on days 2, 9, 16, 23, and 30, and anti-OX40 antibody BMS-986178 IV on days 2, 30, 58, 86, 114, and 142 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-OX40 Antibody BMS 986178; Other: Laboratory Biomarker Analysis; Radiation: Radiation Therapy; Drug: TLR9 Agonist SD-101

INTERVENTIONS:
Biological: Anti-OX40 Antibody BMS 986178 — Given IV, intratumoral
  Other Names: BMS 986178; BMS-986178
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; RADIATION; Radiotherapeutics; radiotherapy; RT; Therapy, Radiation
Drug: TLR9 Agonist SD-101 — Given intratumorally
  Other Names: ISS-ODN SD-101; SD-101

SUMMARY:
This phase I trial studies the side effects and best dose of the anti-OX40 antibody BMS-986178 when given together with the TLR9 agonist SD-101 and radiation therapy in treating patients with low-grade B-cell Non-Hodgkin lymphomas. TLR9 agonist SD-101 may stimulate the immune system in different ways and stop cancer cells from growing. Anti-OX40 antibody is a monoclonal antibody that enhances the activation of T cells, immune cells that are important for fighting tumors Radiation therapy uses high energy x-rays to kill cancer cells and may make them more easily detected by the immune system. Giving TLR9 agonist SD-101 together with anti-OX40 antibody BMS 986178 and radiation therapy may work better in treating patients with low-grade B-cell non-hodgkin lymphomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of TLR9 agonist SD-101 (SD-101) in combination with anti-OX40 antibody BMS 986178 (BMS-986178) and local low-dose radiation in patients with low-grade B-cell lymphoma. Adverse events and grades to be assessed by Common Terminology Criteria for Adverse Events (CTCAE) II. To determine the recommended phase 2 dose (RP2D) of BMS-986178 in combination with intratumoral SD-101 and radiation in patients with low-grade B-cell lymphoma.

SECONDARY OBJECTIVES:

I. To evaluate preliminary efficacy by assessing overall response rate and progression-free survival after treatment with intratumoral SD-101 in combination with BMS-986178 and radiation in patients with low-grade B-cell lymphoma.

OUTLINE: This is a phase I study of the combination of TLR9 agonist SD-101, anti-OX40 antibody BMS 986178, and local low-dose radiation therapy.

Patients receive radiation therapy on days 1-2, TLR9 agonist SD-101 intratumorally on days 2, 9, 16, 23, and 30, and anti-OX40 antibody BMS-986178 intravenously (IV) on days 3, 30, 58, 86, 114, and 142 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed low-grade B-cell lymphoma, excluding gastric MALT lymphoma, high-risk mantle cell lymphoma, and currently transformed lymphoma
* Patients must have at least one site of disease (cervical, axillary, inguinal, or subcutaneous) that is accessible for intratumoral injection of SD-101 (diameter ≥10mm) percutaneously and presents a low risk for complications from direct injections.
* Patients must have at least one site of measurable disease, other than the injection site, which is not included in the radiation field
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count (ANC) >= 1000/mm^3 independent of growth factor support
* Platelets: >= 100,000/mm^3 or >= 50,000/mm^3 if known or suspected bone marrow involvement, independent of transfusion support in either situation
* Hemoglobin: >= 8 g/dL (may be transfused)
* Creatinine: Creatinine clearance > 25 ml/min
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT): =< 3 x upper limit of normal (ULN)
* Bilirubin: =< 1.5 x ULN (except for subjects with Gilbert's Syndrome or of non-hepatic cause)
* Must be at least 4 weeks since treatment with standard or investigational chemotherapy, biochemotherapy, surgery, radiation, cytokine therapy, any monoclonal antibodies or immunotherapy, and recovered from any clinically significant toxicity experienced during treatment
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials; men must agree to not donate sperm during and after the study; for sexually active women of childbearing potential, these restrictions apply for 5 months after the last dose of study drug; for sexually active men, these restrictions apply for 7 months after the last dose of study drug
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at screening, within 24 hours of the first dose of anti-OX40 antibody, and every four weeks while on study treatment; women who are pregnant or breastfeeding are ineligible for this study
* Life expectancy greater than 3 months
* Ability to comply with the treatment schedule
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Currently transformed lymphoma, high-risk mantle cell lymphoma, or gastric MALT lymphoma.
* Need for immediate treatment or cytoreduction.
* No easily accessible site for direct percutaneous injection with low-risk for potential complications.
* Autoimmune disease requiring treatment within the last 5 years including systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, uveitis, or other if clinically significant
* Major surgery within 4 weeks of enrollment, or a wound that has not fully healed
* Vaccinated with live, attenuated vaccines within 4 weeks of enrollment
* Known history of human immunodeficiency virus (HIV) or active hepatitis C virus or active hepatitis B virus infection or any uncontrolled active systemic infection
* Known central nervous system (CNS) lymphoma
* Patients with a history of prior malignancy with the exception of non-melanoma skin cancer, stage 1 prostate cancer that does not require treatment, or other malignancy that has undergone potentially curative therapy with no evidence of disease for the last 2 years and that is deemed by the investigators to be at low risk for recurrence. In situ cancer of any type and noninvasive follicular thyroid neoplasm with papillary-like nuclear features (NIFTP) is not an exclusion, though if surgery or other definitive intervention is planned, it should be completed prior to enrollment.
* History of significant allergic reactions attributed to compounds of similar composition to SD-101 or BMS-986178
* Treatment with an immunosuppressive regimen of corticosteroids or other immunosuppressive medication (e.g., methotrexate, rapamycin) within 30 days of study treatment; Note: patients may take up to 5 mg of prednisone or equivalent daily; topical and inhaled corticosteroids in standard doses are allowed
* Significant cardiovascular disease (i.e. New York Heart Association [NYHA] class 3 congestive heart failure; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty with the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias)
* Pregnant or breast feeding
* Any other medical history, including laboratory results, deemed by the investigator likely to interfere with their participation in the study, or to interfere with the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing Dose-limiting Toxicities (DLT) within 8 weeks of treatment initiation | Up to 8 weeks
  Dose-limiting toxicities (DLTs) as assessed as the following hematologic toxicities (grades per CTCAE) in all participants receiving at least 1 intratumoral (IT) injection of SD-101 and at least 1 dose of BMS-986178 (not including events due to disease progression or definitively unrelated to study drugs):
  * Febrile neutropenia
  * Thrombocytopenia Grade 4 or Grade 3 with bleeding or platelet transfusion
  * Anemia Grade 4
  * Non-hematological toxicity ≥ grade 3, except:
    * Alopecia controlled by medical management
    * Nausea controlled by medical management
    * Grade 3 or 4 electrolyte abnormalities not associated with adverse events, persist < 72 hours, and either spontaneously resolve or respond to intervention.
    * Grade 3 or 4 elevation of amylase or lipase not associated with pancreatitis
    * Grade 3 endocrinopathy
    * Grade 3 infusion reaction returning to ≤ Grade 1 in < 6 hours
    * Grade 3 skin rash not requiring systemic steroid or other immunosuppressive therapy

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 96 weeks
  Overall Response Rate (ORR), assessed as the sum of the complete response (CR) and partial response (PR) rates, as determined by computed tomography (CT) or positron emission tomography (PET)/CT and evaluated per the Lugano classification for low-grade B-cell lymphomas, in all participants receiving at least 1 intratumoral (IT) injection of SD-101 and at least 1 dose of BMS-986178.
  Lugano classification:
  * CR: No detectable disease by CT or PET/CT scan
  * PR: ≥ 50% decrease in size of target lesions
  * No response (NR) / Stable disease (SD): < 50% decrease in size of target lesions
  * Progressive disease (PD): Target lesions larger; clear progression of non-target lesions; or new tumor lesions; new or recurrent bone marrow involvement; splenomegaly + 2 cm or +50%.
  Reported for 24, 48, 72 and 96 weeks.
Progression-Free Survival (PFS) | up to 96 weeks
  Progression-free survival (PFS) as determined for all participants receiving at least 1 intratumoral (IT) injection of SD-101 and at least 1 dose of BMS-986178, from start of treatment to disease progression per the Lugano classification or death from any cause, through 96 weeks. Progression assessed per the Lugano classification. Patients who were last known to be alive and progression-free will be censored at the latest disease assessment.
  Lugano classification:
  * CR: No detectable disease by CT or PET/CT scan
  * PR: ≥ 50% decrease in size of target lesions
  * No response (NR) / Stable disease (SD): < 50% decrease in size of target lesions
  * Progressive disease (PD): Target lesions larger; clear progression of non-target lesions; or new tumor lesions; new or recurrent bone marrow involvement; splenomegaly + 2 cm or +50%.
  Reported for 24, 48, 72 and 96 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Levy, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong WX, Sagiv-Barfi I, Czerwinski DK, Sallets A, Levy R. Neoadjuvant Intratumoral Immunotherapy with TLR9 Activation and Anti-OX40 Antibody Eradicates Metastatic Cancer. Cancer Res. 2022 Apr 1;82(7):1396-1408. doi: 10.1158/0008-5472.CAN-21-1382. PMID 35135810
- [Derived] Mooney KL, Czerwinski DK, Shree T, Frank MJ, Haebe S, Martin BA, Testa S, Levy R, Long SR. Serial FNA allows direct sampling of malignant and infiltrating immune cells in patients with B-cell lymphoma receiving immunotherapy. Cancer Cytopathol. 2022 Mar;130(3):231-237. doi: 10.1002/cncy.22531. Epub 2021 Nov 15. PMID 34780125